CLINICAL TRIAL: NCT05216601
Title: A Phase I, Prospective, Randomized, Open-labeled Study to Evaluate the Safety, Tolerability, and Immunogenicity of Booster Dose With MVC-COV1901 or MVC-COV1901(Beta) SARS-CoV-2 Vaccine in Adults
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of MVC-COV1901 or MVC-COV1901(Beta) Against COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medigen Vaccine Biologics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CT-COV-25
Record Dates: First submitted 2022-01-27; First posted 2022-01-31 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2022-06

CONDITIONS: COVID-19 Vaccine
Keywords: COVID-19 Vaccine
MeSH Terms: interventions — MVC-COV1901 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MVC-COV1901 (Active Comparator): 15 mcg of S-2P protein with adjuvant
  Interventions: Biological: MVC-COV1901
- MVC-COV1901(Beta)-15 (Experimental): 15 mcg of S-2P protein(Beta) with adjuvant
  Interventions: Biological: MVC-COV1901(Beta)-15
- MVC-COV1901(Beta)-25 (Experimental): 25 mcg of S-2P protein(Beta) with adjuvant
  Interventions: Biological: MVC-COV1901(Beta)-25

INTERVENTIONS:
Biological: MVC-COV1901 — Approximately 40 participants who previously completed two (Group A) or three (Group B) doses of MVC-COV1901 will receive 1 doses of MVC-COV1901 at Visit 2 (Day 1) via intramuscular (IM) injection in the deltoid region. Group A and B
  Arms: MVC-COV1901
Biological: MVC-COV1901(Beta)-15 — Approximately 40 participants who previously completed two (Group A) or three (Group B) doses of MVC-COV1901 will receive 1 doses of MVC-COV1901(Beta)-15 at Visit 2 (Day 1) via intramuscular (IM) injection in the deltoid region
  Arms: MVC-COV1901(Beta)-15
Biological: MVC-COV1901(Beta)-25 — Approximately 40 participants who previously completed two (Group A) or three (Group B) doses of MVC-COV1901 will receive 1 doses of MVC-COV1901(Beta)-25 at Visit 2 (Day 1) via intramuscular (IM) injection in the deltoid region
  Arms: MVC-COV1901(Beta)-25

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and immunogenicity of a booster dose of vaccine in participants who are generally healthy or with stable pre-existing health conditions. Study details include:

* The study duration per participant will be approximately 209 days (28 days screening, 1 day vaccination, and 180 days follow-up).
* The treatment duration will be 1 day. -The visit frequency will be 6 on-site visits (1 screening visit, 1 treatment visit, and 4 follow- up visits) and 1 phone visit.

DETAILED DESCRIPTION:
This is a Phase I, prospective, randomized, open-labeled study to evaluate the safety, tolerability, and immunogenicity of a booster vaccination with the MVC-COV1901 or MVC1901(Beta). Approximately 120 participants aged ≥18 and <55 years, who received two or three doses of MVC- COV1901 vaccines, will be enrolled and divided into two groups. Each group will consist of approximately 60 eligible subjects, and for each group the randomization will be stratified based on site to three treatment arms (15 mcg of MVC-COV1901 or 15 mcg or 25 mcg of MVC-COV1901(Beta) in 1:1:1 ratio).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥ 18 years and <55 years at randomization.
2. Healthy adults or adults with pre-existing medical conditions who are in stable condition. A stable medical condition is defined as a disease not requiring significant change in therapy or hospitalization for worsening disease 3 months before enrollment and expected to remain stable for the duration of the study.
3. Documented to have received two or three homologous doses of MVC-COV1901 vaccine, 1st and 2nd doses within 12 weeks, 2nd and 3rd doses between 12~24 weeks (Group B only), and with the latest dose > 84 days prior to randomization, and did not receive any other investigational or approved COVID-19 vaccines.
4. Female participants must:

   1. Be either of non-childbearing potential, i.e. surgically sterilized (defined as having undergone hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy; tubal ligation alone is not considered sufficient) or one year post-menopausal;
   2. Or, if of childbearing potential, be abstinent or agree to use medically effective contraception from 14 days before screening to 30 days following the injection of study intervention. Acceptable forms include:

   i. Implanted hormonal methods of contraception or placement of an intrauterine device or intrauterine system ii. Established use of hormonal methods (injectable, pill, patch or ring) combined with barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository c. Female with childbearing potential must have a negative pregnancy test by this protocol
5. Participant is willing and able to comply with all required study visits and follow-up required
6. Participant, and the participant's legal representative if applicable, must understand the procedures of the study and provide written informed consent.

Exclusion Criteria:

1. Pregnant or breast feeding or plan to become pregnant in 30 days after the administration of study intervention.
2. Employees at the investigator's site, of the Sponsor or delegate (e.g., contract research organization) who are directly involved in the conduct of the study.
3. Currently receiving or received any investigational intervention within 30 days prior to the vaccination of study intervention.
4. Administered any licensed live-attenuated vaccines within 28 days or other licensed non-live- attenuated vaccines within 7 days prior to vaccination of study intervention.
5. Administered any blood product or intravenous immunoglobulin administration within 12 weeks prior to the vaccination of study intervention.
6. Currently receiving or anticipate to receive concomitant immunosuppressive or immune- modifying therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or < 2 weeks of daily receipt of prednisone less than 20 mg or equivalent) within 12 weeks prior to the vaccination of study intervention.
7. Currently receiving or anticipate to receive treatment with tumor necrosis factor (TNF)-α inhibitors, e.g., infliximab, adalimumab, etanercept within 12 weeks prior to the vaccination of study intervention.
8. Major surgery or any radiation therapy within 12 weeks prior to the vaccination of study intervention
9. Immunosuppressive illness or immunodeficient state, including hematologic malignancy, history of solid organ, bone marrow transplantation, or asplenia.
10. A history of malignancy with potential risk for recurrence after curative treatment, or current diagnosis of or treatment for cancer (exceptions are squamous and basal cell carcinomas of the skin and treated uterine cervical carcinoma in situ, at the discretion of the investigator).
11. Bleeding disorder considered a contraindication to intramuscular injection or phlebotomy.
12. Participant with ongoing acute diseases or serious medical conditions which will interfere with adherence to study requirements, or the evaluation of any study endpoint. Acute diseases or serious medical conditions include cardiovascular, pulmonary, hepatic, neurologic, metabolic, renal, psychiatric conditions (e.g., alcoholism, drug abuse, anorexia or severe depression), current severe infections, autoimmune disease, medical history, physical findings, or laboratory abnormality that in the investigators' opinion are not in stable condition and participating in the study could adversely affect the safety of the participant.
13. Documented SARS-CoV-1 or 2 infection prior to the study intervention.
14. Participant with a history of hypersensitivity to any vaccine or a history of allergic disease or reactions likely to be exacerbated by any component of MVC-COV1901 and MVC-COV1901(Beta).
15. Body (oral, rectal, or ear) temperature ≥ 38.0°C or acute illness (not including minor illnesses such as diarrhea or mild upper respiratory tract infection at the discretion of the investigator) within 2 days before the vaccination of study intervention.
16. Any condition that is a contraindication to study intervention based on the judgement of the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events from Day 1 to 29 | Day 1 to Day 29
  To measure the incidence of adverse event from Day 1 to Day 28 after the booster dose.
  * Solicited local adverse events (AEs) (up to 7 days after injection of booster dose) • Solicited systemic AEs (up to 7 days after injection of booster dose)
  * Unsolicited AEs (up to 28 days after injection of booster dose)
  * AE of special interest (AESI)
  * Vaccine-associated enhanced disease (VAED) • Serious adverse event (SAE)
Primary Immunogenicity-1 | Day 1 to Day 29
  To evaluate the immunogenicity in terms of Anti-SARS-CoV-2 neutralizing antibody at Day 29
  • GMT
Primary Immunogenicity-2 | Day 1 to Day 29
  To evaluate the immunogenicity in terms of Anti-SARS-CoV-2 neutralizing antibody at Day 29
  • GMT ratio

SECONDARY OUTCOMES:
Incidence of Adverse Events from Day 1 to 181 | Day 1 to Day 181
  To measure the incidence of adverse event throughout the whole study period.
  * ≥ Grade 3 AE
  * AESI
  * VAED
  * SAE
Secondary Immunogenicity (Humoral)-1 | Day 1 to Day 181
  To evaluate the immunogenicity in terms of Anti-spike IgG
  • GMT
Secondary Immunogenicity (Humoral)-2 | Day 1 to Day 181
  To evaluate the immunogenicity in terms of Anti-spike IgG
  • GMT Ratio
Secondary Immunogenicity (Cellular) | Day 1 to Day 91
  To evaluate the cellular immunology by Enzyme-linked immunoSpot assay (ELISpot)

OTHER OUTCOMES:
Exploratory Immunogenicity-1 | Day 1 to Day 29
  To evaluate the immunogenicity in terms of neutralizing antibody titers against the Variants of Concern (VoCs)
  • GMT
Exploratory Immunogenicity-2 | Day 1 to Day 29
  To evaluate the immunogenicity in terms of neutralizing antibody titers against the Variants of Concern (VoCs)
  • GMT ratio

CONTACTS AND LOCATIONS:
Overall Officials: Allen Lien, MD Dr.Ph, Study Director — Medigen Vaccine Biologics
Locations (2):
- Taiwan (2):
  - Taipei Medical University Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No